CLINICAL TRIAL: NCT05215574
Title: A Phase 1 Dose Escalation/Dose Finding Study of NGM831 as Monotherapy and in Combination With Pembrolizumab or Pembrolizumab and NGM438 in Advanced or Metastatic Solid Tumors
Brief Title: Study of NGM831 as Monotherapy and in Combination With Pembrolizumab or Pembrolizumab and NGM438 in Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 831-IO-101; KEYNOTE-E13 (Other: MK-3475-E13 Merck Sharp & Dohme LLC.)
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Cancer; Breast Cancer; Gastric Cancer; Non-small Cell Lung Cancer; Cervical Cancer; Endocervical Cancer; Squamous Cell Carcinoma of Head and Neck; Bladder Urothelial Cancer; Colorectal Carcinoma; Esophageal Cancer; Ovarian Cancer; Renal Cell Carcinoma; Prostate Cancer; Melanoma; Mesothelioma; Cholangiocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Breast Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Esophageal Neoplasms; Ovarian Neoplasms; Carcinoma, Renal Cell; Prostatic Neoplasms; Melanoma; Mesothelioma; Cholangiocarcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NGM831 Monotherapy Dose Escalation (Experimental): Part 1a Single Agent Dose Escalation
  Interventions: Drug: NGM831
- NGM831 combination dose finding with pembrolizumab (KEYTRUDA®) (Experimental): Part 1b NGM831 plus pembrolizumab (KEYTRUDA®)
  Interventions: Drug: NGM831 plus pembrolizumab (KEYTRUDA®)
- NGM831 and NGM438 Combination Dose Finding with pembrolizumab (KEYTRUDA®) (Experimental): Part 1c NGM831 and NGM438 plus pembrolizumab (KEYTRUDA®)
  Interventions: Drug: NGM831 and NGM438 plus pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Drug: NGM831 — Drug: NGM831 NGM831 is given intravenously (IV) every 3 weeks in a 21 day cycle. Multiple dose levels will be evaluated.
  Arms: NGM831 Monotherapy Dose Escalation
Drug: NGM831 plus pembrolizumab (KEYTRUDA®) — Drug: NGM831 NGM831 is given intravenously (IV) every 3 weeks in a 21day cycle. Multiple dose levels will be evaluated.
  Drug: pembrolizumab (KEYTRUDA®) pembrolizumab (KEYTRUDA®) will be administered intravenously (IV) every 3 weeks in a 21day cycle.
  Arms: NGM831 combination dose finding with pembrolizumab (KEYTRUDA®)
Drug: NGM831 and NGM438 plus pembrolizumab (KEYTRUDA®) — Drug: NGM831 NGM831 is given intravenously (IV) every 3 weeks in a 21-day cycle. Multiple dose levels will be evaluated.
  Drug: NGM438 NGM438 is given intravenously (IV) every 3 weeks in a 21-day cycle. Multiple dose levels will be evaluated.
  Drug: pembrolizumab (KEYTRUDA®) pembrolizumab (KEYTRUDA®) will be administered intravenously (IV) every 3 weeks in a 21-day cycle.
  Arms: NGM831 and NGM438 Combination Dose Finding with pembrolizumab (KEYTRUDA®)

SUMMARY:
Study of NGM831 as Monotherapy and in Combination with Pembrolizumab or Pembrolizumab and NGM438 in Advanced or Metastatic Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced or metastatic solid tumor malignancy.
* Adequate bone marrow, kidney and liver function
* Performance status of 0 or 1.
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade 1 except for AEs not constituting a safety risk by Investigator judgement.

Exclusion Criteria:

* Prior treatment targeting ILT3.
* Prior treatment targeting LAIR1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose-limiting Toxicities | Baseline up to 21 Days
  A DLT is defined as an AE that meets at least one of the criteria listed in protocol, according to National Cancer Institute (NCI) common terminology criteria for AE (CTCAE) version 5.0 and is considered by the Investigator to be clinically relevant and attributed to the study treatment during the first 21 days after the first dose of study treatment.
Incidence of Adverse Events | Baseline up to Approximately 24 months
  Number of patients with treatment-emergent adverse events (AEs) An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of patients who experience at least one AE will be presented.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of NGM831 | Baseline up to approximately 9 weeks
  Cmax is defined as the observed maximum serum concentration post drug administration.
  Will be measured for Cycle 1 and Cycle 3.
Time to Maximum Observed Serum Concentration (Tmax) of NGM831 | Baseline up to approximately 9 weeks
  Tmax is defined as the time to reach the observed maximum serum concentration (Cmax) post drug administration.
  Will be measured for Cycle 1 and Cycle 3.
Area Under the Concentration Time Curve of the dosing interval (AUC) of Serum NGM831 | Baseline up to approximately 9 weeks
  AUC is defined as area under the concentration time curve of the dosing interval post drug administration.
  Will be calculated for Cycle 1 and Cycle 3.
Maximum Observed Serum Concentration (Cmax) of NGM438 | Baseline up to approximately 9 weeks
  Cmax is defined as the observed maximum serum concentration post drug administration.Will be measured for Cycle 1 and Cycle 3.
Time to Maximum Observed Serum Concentration (Tmax) of NGM438. | Baseline up to approximately 9 weeks
  Tmax is defined as the time to reach the observed maximum serum concentration (Cmax) post drug administration.
  Will be measured for Cycle 1 and Cycle 3.
Area Under the Concentration Time Curve of the dosing interval (AUC) of Serum NGM438 | Baseline up to approximately 9 weeks
  AUC is defined as area under the concentration time curve of the dosing interval post drug administration.
  Will be calculated for Cycle 1 and Cycle 3.
Anti-drug Antibodies (ADA) Against NGM831 | Baseline up to approximately 24 months
  Incidence and titers of anti-drug antibodies (ADA) against NGM831. Will be measured on Day 1 of each cycle.
Anti-drug Antibodies (ADA) Against NGM438 | Baseline up to approximately 24 months
  Incidence and titers of anti-drug antibodies (ADA) against NGM438. Will be measured on Day 1 of each cycle.
Neutralizing antibodies (nAb) against NGM831 | Baseline up to approximately 24 months
  Incidence and titers of neutralizing antibodies (nAb) against NGM831. Will be measured on Day 1 of each cycle.
Neutralizing antibodies (nAb) against NGM438 | Baseline up to approximately 24 months
  Incidence and titers of neutralizing antibodies (nAb) against NGM438. Will be measured on Day 1 of each cycle.
Number of Patients with Objective Responses | Baseline up to approximately 24 months
  Objective Response Rate is defined as the proportion of patients who achieve a confirmed complete response (CR) or partial response (PR) divided by the total number of evaluable patients per RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - NGM Clinical Study Site, Gilbert, Arizona
  - NGM Clinical Study Site, Los Angeles, California
  - NGM Clinical Study Site, Sarasota, Florida
  - NGM Clinical Study Site, Tampa, Florida
  - NGM Clinical Study Site, Grand Rapids, Michigan
  - NGM Clinical Study Site, New York, New York
  - NGM Clinical Study Site, Oklahoma City, Oklahoma
  - NGM Clinical Study Site, Austin, Texas
  - NGM Clinical Study Site, Houston, Texas